CLINICAL TRIAL: NCT05090293
Title: Optimizing Weight Loss Outcomes Through Body Image Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Martin Binks, Associate Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTUIRB2021-470
Record Dates: First submitted 2021-09-21; First posted 2021-10-22 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (LI) (Active Comparator): Participants will receive a standard, 12-week, group-delivered cognitive behavioral lifestyle intervention for weight loss.
  Interventions: Behavioral: Lifestyle Intervention (LI)
- Lifestyle Intervention with Body Image Treatment (LIBI) (Experimental): Participants will receive a standard, 12-week, group-delivered cognitive behavioral lifestyle intervention for weight loss supplemented with a novel body image intervention designed to address body image issues in the context of weight loss.
  Interventions: Behavioral: Experimental: Lifestyle Intervention with Body Image Treatment (LIBI)

INTERVENTIONS:
Behavioral: Experimental: Lifestyle Intervention with Body Image Treatment (LIBI) — A body image protocol designed to improve outcomes in a group-delivered multidisciplinary weight loss program by addressing body acceptance within a context of positive behavior change and utilizing existing body discomfort and re-purposing it as an agent of motivation.
  Arms: Lifestyle Intervention with Body Image Treatment (LIBI)
Behavioral: Lifestyle Intervention (LI) — A multidisciplinary, group-delivered, multidisciplinary weight loss program addressing various lifestyle factors impacting weight loss.
  Arms: Lifestyle Intervention (LI)

SUMMARY:
The study will examine if a standard group-delivered cognitive behavioral lifestyle intervention for weight loss can be improved via the incorporation of a novel body image intervention designed to address body image and improve weight loss outcomes in a sample of women with overweight/obesity.

DETAILED DESCRIPTION:
Weight loss is associated with improved morbidity and mortality in people with overweight/obesity. Lifestyle-focused interventions reliably produce modest weight loss. While some comprehensive multidisciplinary weight management interventions include behavioral and psychosocial aspects of behavior change, including brief body image education, few have focused substantially on body image as a potentially salient influence on motivation and/or successful outcomes. Body image is an individual's perception of their physical self. A common psychosocial correlate of obesity is body dissatisfaction, and research has shown that individuals with obesity are more often dissatisfied with their bodies than individuals without obesity. Multiple studies suggest that improving body image might enhance eating self-regulation during weight management interventions and engagement in physical activity. Additionally, negative body image has been associated with detrimental health outcomes, such as emotional eating and avoidance of physical activity. Although body image has been addressed in the context of obesity and weight management, it is often done in a cursory manner. To date, no weight loss programs have attempted to develop a novel body image intervention that specifically targets the necessary dichotomy between body acceptance and expectable desire for body changes in a weight loss program. As such, the investigators will examine if a standard group-delivered cognitive behavioral lifestyle intervention for weight loss can be improved via the incorporation of a novel body image intervention designed to address body image and improve weight loss outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 and older
* Sex: Female
* BMI of 25 kg/m2 or greater

Exclusion Criteria:

* Participants unable or unwilling to provide informed consent
* Participants who are pregnant or planning to become pregnant over the next 4 months
* Participants who are breastfeeding or planning to breastfeed over the next 4 months
* Participants who have received a diagnosis of diabetes (type I or II)
* Participants who been told NOT to lose weight or exercise for any reason by a healthcare provider
* Participants who currently have psychiatric illnesses (e.g., Psychosis, schizophrenia, bipolar disorder or severe depression/anxiety)
* Participants who currently have persistent suicidal thoughts or have attempted suicide in the last year
* Participants with a history of diagnosed eating disorders such as bulimia nervosa or anorexia nervosa.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
Comparison of Weight | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in weight loss
Comparison of Body Fat Mass | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in body fat mass
Comparison of Blood Pressure | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in systolic blood pressure
Comparison of Blood Pressure | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in diastolic blood pressure
Comparison of Blood Pressure | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in resting heart rate
Comparison of Physical Activity Engagement | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Increase in self-reported physical activity engagement
Comparison of Health Related Quality of Life | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Increase in self-reported health related quality of life
Comparison of Body Image | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in attitudinal and perceptual body image

SECONDARY OUTCOMES:
Comparison of Interoceptive Awareness | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in the ability to identify and respond appropriately to internal bodily signals
Comparison of General Self-Efficacy | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in self-perception of ability and competence to perform effectively across different tasks and situations
Comparison of Dieting Self-Efficacy | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in self-perception of adequately responding to scenario-based eating temptations
Comparison of Exercising Self-Efficacy | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in self-perception of belief in ability to continue exercising despite setbacks
Comparison of Fear of Negative Evaluation | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in self-reported apprehension about negative evaluations by others
Comparison of Motivation to Engage in Physical Activity | Baseline (pre-intervention) and 14 weeks (post-intervention)
  Changes in self-reported motivation to engage in physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Martin Binks, Ph.D., Principal Investigator — Texas Tech University- Department of Nutritional Sciences
Locations (2):
- United States (2):
  - Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas
  - Nutrition & Metabolic Health Initiative, Lubbock, Texas